CLINICAL TRIAL: NCT07084519
Title: Randomized Controlled Trial of Postmastectomy Hypofractionated Radiotherapy Versus Conventional Fractionated Radiotherapy in Breast Cancer Patients Undergoing Prosthetic Breast Reconstruction
Brief Title: Hypofractionated vs Conventional RT After Prosthetic Breast Reconstruction
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor of radiation oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5419
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Reconstruction; Radiation Oncology
Keywords: breast cancer; prosthetic breast reconstruction; hypofractionated radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFRT group (Experimental): 43.5 Gy in 15 fractions (2.9 Gy/fraction, 3 weeks)
  Interventions: Radiation: hypofractionated radiotherapy
- CFRT group (Other): 50 Gy in 25 fractions, 2 Gy/fraction, 5 weeks
  Interventions: Radiation: conventional fractionated radiotherapy

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — 43.5 Gy in 15 fractions (2.9 Gy/fraction, 3 weeks)
  Arms: HFRT group
Radiation: conventional fractionated radiotherapy — 50 Gy in 25 fractions, 2 Gy/fraction, 5 weeks
  Arms: CFRT group

SUMMARY:
This study investigates the safety and efficacy of hypofractionated radiotherapy (HFRT) versus conventional fractionated radiotherapy (CFRT) in breast cancer patients undergoing total mastectomy with prosthetic reconstruction.

Study Design Population: Patients with high-risk breast cancer after mastectomy and immediate implant reconstruction.

Intervention:

HFRT Arm: 43.5 Gy in 15 fractions (2.9 Gy/fraction, 3 weeks). Control Arm: CFRT (50 Gy in 25 fractions, 2 Gy/fraction, 5 weeks). Endpoints Primary: Reconstruction failure rate (e.g., implant removal, capsular contracture)

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-75 years
* Karnofsky Performance Status ≥60
* Histopathologically confirmed invasive breast adenocarcinoma
* Total mastectomy [with or without nipple-areolar complex preservation] + axillary dissection/sentinel lymph node biopsy + implant/expander placement R0 resection with negative margins
* pT3 or N2-3 disease; or pT1-2N1
* No distant metastasis
* Completed standard neoadjuvant/adjuvant chemotherapy cycles
* ≤8 weeks post-chemotherapy or ≤12 weeks post-surgery if no chemotherapy
* Signed informed consent

Exclusion Criteria:

* Prior radiotherapy to chest wall or nodal regions
* Pregnancy or lactation
* T4 stage disease
* Pre-radiotherapy local/regional/distant metastasis
* Grade ≥3 implant-related adverse events irreversible before radiotherapy
* Bilateral breast cancer requiring bilateral radiotherapy
* Concurrent/secondary malignancy with disease-free interval <5 years [except non-melanoma skin cancer, papillary/follicular thyroid cancer, or cervical carcinoma in situ]
* Active collagen vascular disease, e.g., SLE, scleroderma
* Uncontrolled comorbidities: acute cardiovascular disease, substance abuse, or psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Reconstruction Failure Rate | 2 year
  implant removal, capsular contracture ≥ Baker grade III

SECONDARY OUTCOMES:
Other Implant-Related Adverse Events | 2 year
  infection, skin necrosis, implant exposure
Radiation-Related Toxicities | 2 year
  grade ≥3 dermatitis, pneumonitis, lymphedema
DFS | 5 year
  Disease-Free Survival
OS | 5 year
  Overall Survival
LRR | 5 year
  Locoregional Recurrence Rate
DM | 5 year
  Distant Metastasis Rate
Cosmetic Outcome Assessed by Harvard Breast Cosmesis Scale (Physician-Rated) | 1 year
  Physicians will assess cosmetic outcome using the Harvard Breast Cosmesis Scale.
  Unit of Measure: Score on Harvard Breast Cosmesis Scale Scale Information: Score range from 1 (Excellent) to 4 (Poor). Higher scores indicate worse cosmetic outcomes.
Patient-Reported Cosmetic Outcome | 1 year
  Description: Patients will self-assess cosmetic outcome using a 4-point Likert scale.
  Unit of Measure: Score on 4-point Likert scale. Scale Information: Score range from 1 (Excellent) to 4 (Poor). Higher scores indicate worse perceived outcome.
Quality of Life Assessed by EORTC QLQ-C30 Global Health Status Score | Baseline, 6 months, and 12 months after treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) will be used to evaluate patients' global health status and overall quality of life.
  Unit of Measure: Score on a scale Scale Information: Score ranges from 0 to 100; higher scores indicate better global health status.
Quality of Life Assessed by EORTC QLQ-BR23 Breast Cancer Module | Baseline, 6 months, and 12 months after treatment
  The EORTC Quality of Life Questionnaire Breast Cancer Module (EORTC QLQ-BR23) will be used to assess breast cancer-specific quality of life.
  Unit of Measure: Score on a scale Scale Information: Score ranges from 0 to 100. For functional scales, higher scores indicate better function; for symptom scales, higher scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Province, China

IPD SHARING:
Plan to Share IPD: No
IPD includes sensitive participant information. Premature sharing could compromise publication opportunities or patent filings.